CLINICAL TRIAL: NCT06669416
Title: Effects of Patient Education and Self-Management in Cancer Patients Who Experience Chemotherapy-Induced Taste Alterations
Brief Title: Taste Alterations Study
Acronym: TAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00120499
Record Dates: First submitted 2024-10-25; First posted 2024-11-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chemotherapy Side Effects; Taste, Altered
Keywords: self-management; cluster randomized control trial
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Intervention Model Description: Treatment/Control (usual care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/Usual Care (No Intervention): Chemotherapy infusion clinics deliver infusion services based on the American Society of Clinical Oncology (ASCO) Quality Oncology Practice Initiative (QOPI) Chemotherapy Administration Safety Standards (2020) including standard toxicity screening and providing standard chemotherapy patient education with general information for managing nausea and other gastrointestinal side effects and nutrition tips. Usual care patients will be supplemented with a single-item question to evaluate taste alteration severity and to gather information about what they are doing and their diet intake.
- Treatment - TA Self-monitoring and Self-management (Experimental): The nurse-led intervention involves using a valid/reliable TA assessment tool (Chemotherapy-induced Taste Alterations Scale (CiTAS) and teaching the patient to use the assessments and the evidence-based Patient Education Sheet to select assessment-driven interventions to manage TA symptoms. Data is collected about the specific actions prescribed in the teaching tool to identify which interventions were used and their overall impact.
  Interventions: Behavioral: Taste Alteration Self-Assessment; Behavioral: Taste Alternation Self-Management

INTERVENTIONS:
Behavioral: Taste Alteration Self-Assessment — The nurse-led intervention involves using a valid/reliable TA assessment tool (Chemotherapy-induced Taste Alterations Scale (CiTAS) and teaching the patient to select assessment-driven interventions to manage TA symptoms.
  Arms: Treatment - TA Self-monitoring and Self-management
Behavioral: Taste Alternation Self-Management — The nurse-led intervention involves teaching the patient to use the assessments and the evidence-based Patient Education Sheet to select assessment-driven interventions to manage their symptoms. Data will be collected about the specific actions prescribed in the teaching tool and to identify which interventions were used and their overall impact.
  Arms: Treatment - TA Self-monitoring and Self-management

SUMMARY:
The main questions it aims to answer are:

1. Does completing a standard assessment increase the detection of chemotherapy induced taste changes compared with usual care (no assessment)? What TA are experienced? Are there any patterns in TA symptom occurrence based on age, sex, race/ethnicity, cancer type, chemotherapy agent, etc.
2. Do patients take action to deal with the TA? What strategies are used? Do patients in the intervention group use the assessments to select interventions?
3. Do the interventions lessen TA symptoms and maintain food intake? Is the treatment (in-depth assessment and education) more effective in lessening the intensity of TA than usual care? Which level of assessment is needed to support symptom management to reduce symptom severity?

Participants will:

Complete baseline assessment before starting their initial chemotherapy infusion (all patients) Participate in baseline patient education based on assigned intervention (usual care vs. treatment) Engage in TA management between chemotherapy infusion clinic visits based on education Visit the clinic for chemotherapy infusions as scheduled; Complete TA assessments and reporting based on intervention; Work with nurse coaches to answer questions and help with the intervention.

Complete study data collection on the 4th chemotherapy cycle (but continue intervention) Complete final data collection at 6 months

DETAILED DESCRIPTION:
BACKGROUND/RATIONALE: Chemotherapy-induced taste alteration (TA) is a common problem for cancer patients with reported prevalence ranging from 35% to 69%. TA systems are associated with decreased dietary intake, malnutrition, and decreased quality of life with no known treatment. Researchers have demonstrated that breast cancer patients were able to control TA with the use of patient self-monitoring and self-management strategies, but these strategies are relatively untested. Research is needed to confirm the effectiveness of this nurse-led intervention when delivered by clinicians with a heterogeneous patient population.

PURPOSE To increase our understanding of the patient experience with TA during chemotherapy and test if adding steps to assess and lessen taste alterations works better than usual care. The infusion clinics will be randomly assigned and trained to provide usual care or usual care with added strategies. Patients receive care method based on clinic assignment (control/treatment). The study does not involve the use of experimental drugs, devices, or procedure.

METHOD: This prospective cluster randomized controlled trial (RCT) is designed to enroll consenting adult cancer patients (n=50/clinic x 8 clinics; N=400) who initiate chemotherapy to evaluate the effect of a nurse-led intervention to engage patients in assessing and self-managing taste alterations (TA) during the first (4) chemotherapy cycles with six months.

INTERVENTION: The nurse-led intervention involves using a single item TA assessment question and an intervention tracking process to evaluate change in outcomes for both groups. The intervention involves using a more extensive valid/reliable assessment tool (Chemotherapy-induced Taste Alterations Scale (CiTAS) teaching the patient to use the findings and the evidence-based Patient Education sheet to select assessment-driven interventions to manage TA symptoms.

OUTCOMES: TA severity (single item and scale); Interventions Used; Patient-reported Effect; Dietary Intake, and BMI.

This study will advance the science by designing and testing the effectiveness of a nurse-led intervention to support infusion clinic patients in TA self-monitoring and management for a heterogenous patient populations beyond breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of cancer with types limited to the top cancer types [Note: Cancer types that are rare will be excluded]
* Initiating chemotherapy (first day/first cycle) at participating clinics
* English speaking/reading (without an interpreter)

Exclusion Criteria:

* Substitute decision-maker (activated)
* History of head/neck cancer or irradiation
* Known genetic/metabolic disorder impacting taste (preexisting dysgeusia)
* Known eating disorder
* Receiving enteral or parenteral nutrition (special nutritional needs)
* Pregnant women (unique needs)
* Patients with medical orders for end of life/hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Taste Alteration Severity | Through study completion, an average of 6 months.
  A single item question with ordinal rating will be used to confirm taste alterations and evaluate severity of TA (control) The CiTAS tool (18 item ordinal rating tool) will be used to confirm taste alterations and evaluate severity of TA (treatment)
Body mass index (BMI) | Through study completion, an average of 6 months.
  BMI is measured to monitor for changes in weight relative to height; It is used to monitor for changes in weight that may indicate that patient is experiencing weight loss during chemotherapy treatment.
Dietary intake | Through study completion, an average of 6 months.
  All patients will be asked to report number of meals/day, number of snacks/day, and number of supplements per day as an estimate of food intake during chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mary L Hook, PhD, RN, Principal Investigator — Aurora Sinai Medical Center
Locations (1):
- Advocate Illinois Masonic Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kano T, Kanda K. Development and validation of a chemotherapy-induced taste alteration scale. Oncol Nurs Forum. 2013 Mar;40(2):E79-85. doi: 10.1188/13.ONF.E79-E85. PMID 23448748
- [Background] Kinjo T, Kanda K, Fujimoto K. Effects of a self-monitoring intervention in breast cancer patients suffering from taste alterations induced by chemotherapy: A randomized, parallel-group controlled trial. Eur J Oncol Nurs. 2021 Jun;52:101956. doi: 10.1016/j.ejon.2021.101956. Epub 2021 Apr 14. PMID 33940487
- [Background] Asano S, Sawatari H, Mentani H, Shimada Y, Takahashi M, Fudano K, Sasaki K, Niitani M, Tanabe K, Kataoka T. Taste Disorders: Effect of Education in Patients With Breast Cancer Receiving Chemotherapy. Clin J Oncol Nurs. 2020 Jun 1;24(3):265-271. doi: 10.1188/20.CJON.265-271. PMID 32441675
- [Background] Barlow LA. The sense of taste: Development, regeneration, and dysfunction. WIREs Mech Dis. 2022 May;14(3):e1547. doi: 10.1002/wsbm.1547. Epub 2021 Nov 30. PMID 34850604
- [Background] Braud A, Boucher Y. Taste disorder's management: a systematic review. Clin Oral Investig. 2020 Jun;24(6):1889-1908. doi: 10.1007/s00784-020-03299-0. Epub 2020 May 8. PMID 32385655
- [Background] Buttiron Webber T, Briata IM, DeCensi A, Cevasco I, Paleari L. Taste and Smell Disorders in Cancer Treatment: Results from an Integrative Rapid Systematic Review. Int J Mol Sci. 2023 Jan 28;24(3):2538. doi: 10.3390/ijms24032538. PMID 36768861
- [Background] Joseph PV, Nolden A, Kober KM, Paul SM, Cooper BA, Conley YP, Hammer MJ, Wright F, Levine JD, Miaskowski C. Fatigue, Stress, and Functional Status are Associated With Taste Changes in Oncology Patients Receiving Chemotherapy. J Pain Symptom Manage. 2021 Aug;62(2):373-382.e2. doi: 10.1016/j.jpainsymman.2020.11.029. Epub 2020 Nov 28. PMID 33259906
- [Background] von Grundherr J, Koch B, Grimm D, Salchow J, Valentini L, Hummel T, Bokemeyer C, Stein A, Mann J. Impact of taste and smell training on taste disorders during chemotherapy - TASTE trial. Cancer Manag Res. 2019 May 16;11:4493-4504. doi: 10.2147/CMAR.S188903. eCollection 2019. PMID 31191011
- [Background] Kumbargere Nagraj S, George RP, Shetty N, Levenson D, Ferraiolo DM, Shrestha A. Interventions for managing taste disturbances. Cochrane Database Syst Rev. 2017 Dec 20;12(12):CD010470. doi: 10.1002/14651858.CD010470.pub3. PMID 29260510